CLINICAL TRIAL: NCT01151735
Title: Randomized, Double-blind, Placebo-controlled, Dose-finding Study to Determine the Efficacy of 1000u, and 1500u of C1-INH Compared to Placebo at the Time of Prodromal Symptoms in Preventing an Acute HAE Exacerbation.
Brief Title: C1-INH Compared to Placebo at the Time of Prodromal Symptoms for Hereditary Angioedema (HAE) Exacerbation
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PennState would not allow the study to move forward
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Timothy Craig, Principal Investigator, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB#33225
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Hereditary Angioedema
Keywords: Angioedema; Hereditary Diseases; Orphan Disease; HAE
MeSH Terms: conditions — Angioedemas, Hereditary; Angioedema; Genetic Diseases, Inborn; Rare Diseases | interventions — Complement C1; Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- C-1-esterase inhibitor 1000 units (Active Comparator): 1000 units of C-1-esterase inhibitor given at time of prodromal symptoms
  Interventions: Drug: C-1-esterase
- 1500 units of C-1-esterase inhibitor (Active Comparator): treatment with 1500 units of C-1-esterase inhibitor IV at the time of prodromal symptoms to decrease risk of exacerbation of HAE
  Interventions: Drug: C-1-esterase
- placebo injection (Placebo Comparator): placebo injection given for prodromal symptoms as double blinded therapy
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: C-1-esterase — 1000 units of C-1-esterase inhibitor
  Other Names: low dose intervention
  Arms: C-1-esterase inhibitor 1000 units
Drug: C-1-esterase — 1500 units of C-1-esterase inhibitor
  Other Names: high dose intervention
  Arms: 1500 units of C-1-esterase inhibitor
Drug: placebo — placebo
  Other Names: placebo arm
  Arms: placebo injection

SUMMARY:
The study hypothesis is that treatment of Hereditary Angioedema at the time of prodromal symptoms will decrease morbidity associated with the disease

DETAILED DESCRIPTION:
Section 3 Study Design and Methods:

Our proposal is to perform a randomized double-blind, three-arm, three-way cross-over study in which subjects with HAE would be placed into one of three different treatment groups based on computer randomization. Subjects will be randomized to receive placebo, 1000 units, or 1500 units of C1-INH at the onset of prodromal symptoms although they would be blinded to which one they were receiving. Randomization will be to one of the two doses or placebo and the sequence of further treatments will be determined randomly in a double-blinded fashion by a person who is not involved in the study. The randomized drug will be available 24 hours and 7 days a week. They would have to come to the study office to receive the blinded drug, and would need to seek treatment within 6 hours of the onset of the prodrome. Following the blinded treatment, the subject would need to be observed for at least 30 minutes. If a subject develops an acute HAE exacerbation in any of the three treatment periods, they would have access to 20 units/kg of open label C1-INH for acute treatment also received at the study office, and the time from onset of symptoms of an acute attack until the time the subject sought open-label treatment could not exceed 12 hours. Following open label rescue, the subject would need to be observed for at least 1 hour or until symptoms started to improve. The subject would also be expected to complete a symptom diary card over the next 24 hours after receiving open-label C1-INH to monitor severity and duration of symptoms (24 Hour Prodrome/Open-Label Diary Appendix IV) associated with the acute attack. The number, duration, and severity of acute HAE attacks would be compared for each treatment period. Each treatment period would last 16 weeks so each subject would be studied for a total of 48 weeks. Because safety has been established when C1-INH is used every third day with prophylaxis therapy, and patients may receive C1-INH for an attack without limits on the closeness of the attacks, our patients in this study may be retreated for prodromal symptoms as they require it, but not more than every other day since prodromes may precede the swelling and abdominal pain by up to 2 days.

Thrombosis has been identified with C1-INH, but only in neonates who were premature and at much higher doses than 1500 units every third day. Cinryze, also a C1-INH, is FDA approved for 1000 units every third day for prophylaxis. The dosing used in our study reflects the FDA approval dosing for Berinert, which is 20 units per kg for acute therapy, so that most patients will receive 1000 to 2500 units of C1-inh whenever they have an attack without day restrictions between dosing. The dosage approved by the FDA is 20 units per kg for Berinert and 1000 units total dose for Cinryze. The dose used in our study approximates these doses, but is not an FDA approved dose. There are no limits on how often Berinert can be dosed for acute attacks.

Figure IV outlines our treatment protocol.

Figure IV: Three-arm, randomized, cross-over, double-blind, placebo-controlled trial to determine effect of treating prodromal symptoms with C1-INH infusions of 1000 units, or 1500 units versus placebo. The sequence is random and double-blinded.

ELIGIBILITY:
Inclusion Criteria:

1. Documented HAE type 1 or 2 by C4 level and C1-INH level or function.
2. Able to read, understand, and sign informed consent.
3. Above the age of 12 years.
4. Willing to complete daily diary.
5. Have at least 1 HAE exacerbations per month averaged over the last 6 months.
6. Prodromal symptoms will not be an inclusion or exclusion since if used it would bias our ability to determine specificity and sensitivity of prodromal symptoms.
7. Present for treatment within 6 hours of onset of prodromal symptoms.
8. Treatment for an acute attack can be given at any time without restriction.

Exclusion Criteria:

1. Inability to read English.
2. Prior adverse effects to C1-INH.
3. Participation in alternate investigational drug trial.
4. Diabetes, neurologic diseases, cardiac diseases, dermatologic diseases that may have associated symptoms that mimic prodromal symptoms.
5. Inability to withdraw from androgens or C1-INH prophylaxis.
6. Pregnant or breast feeding mothers.
7. Prisoners or other institutionalized individuals.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
percentage of full blown HAE attacks occurring within 24 hours following treatment at the prodromal | 24 hours
  To compare the percentage of full blown HAE attacks occurring within 24 hours following treatment at the prodromal stage of an attack using placebo or one of two doses of C1-INH.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lunn, DO, Principal Investigator — Penn State University